CLINICAL TRIAL: NCT04595812
Title: Comparing Preoperative Vaginal Misoprostol, Intraoperative Oxytocin Infusion, Intravenous Carbetocin and Pericervical Hemostatic Tourniquet in Reducing Blood Loss During Abdominal Myomectomy, a Randomized Controlled Trial
Brief Title: Methods to Reduce Blood Loss in Abdominal Myomectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Hany Mohamed, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Reduce bleeding in myomectomy
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Abdominal Myomectomy; Blood Loss
Keywords: misoprostol; oxytocin; carbetocin; tourniquet
MeSH Terms: conditions — Hemorrhage | interventions — Misoprostol; Oxytocin; carbetocin

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Misoprostol group (Active Comparator): receive two tablets of 200µg misoprostol (Pfizer Limited, United Kingdom) administered into the posterior fornix of the vagina 1 hour before the onset of surgery
  Interventions: Drug: Misoprostol 200mcg Tab vaginal
- Oxytocin group (Active Comparator): After induction of general anaesthesia and immediately prior to the operation, an infusion of 30 IU oxytocin in 500 ml normal saline at a rate of 120 ml/h will be started during myomectomy.
  Interventions: Drug: Oxytocin
- Carbetocin group (Experimental): receive 100 μg IV Carbetocin (1ml) [Pabal, Ferring (UK)] in 5 ml saline over 1 minute just before skin incision
  Interventions: Drug: Carbetocin
- pericervical tourniquet group (Active Comparator): pericervical tourniquet using a Foley catheter size 18, which will be firmly tied at the level of the cervico-isthmic junction of the uterus before the uterine incision.
  Interventions: Procedure: pericervical hemostatic tourniquet

INTERVENTIONS:
Drug: Misoprostol 200mcg Tab vaginal — 2 tablets vaginally 1 hour before surgery
  Other Names: cytotec
  Arms: Misoprostol group
Drug: Oxytocin — 30 IU oxytocin in 500 ml normal saline at a rate of 120 ml/h
  Arms: Oxytocin group
Drug: Carbetocin — 100 μg IV Carbetocin (1ml) in 5 ml saline over 1 minute
  Other Names: Pabal, Ferring (UK)
  Arms: Carbetocin group
Procedure: pericervical hemostatic tourniquet — a Foley catheter size 18, which will be firmly tied at the level of the cervico-isthmic junction of the uterus before the uterine incision,The time of tourniquet administration will be recorded, and will be released not later than 45 minutes after its application. For those requiring multiple applications, the tourniquet will be reapplied after a period of at least 15 minutes.
  Arms: pericervical tourniquet group

SUMMARY:
The aim of the study is to compare the effectiveness of a single preoperative dose of vaginal misoprostol, intraoperative oxytocin infusion, IV carbetocin and pericervical tourniquet for the reduction of blood loss during of abdominal myomectomy.

DETAILED DESCRIPTION:
Uterine leiomyomas (fibroids) are the most common benign tumours among women. Fibroids are found in approximately 20% of women over 35 years of age. They are mostly asymptomatic, but in 20-50% of patients, fibroids may cause problems such as heavy menstrual bleeding, anaemia, pelvic pain and pressure,symptoms from extrinsic compression of the colorectal and urinary tract,recurrent abortion and infertility. Surgery is indicated for symptomatic uterine leiomyomas; hysterectomy for women who have completed childbearing (women > 40 years old), and myomectomy for women <40 years old who wish to preserve uterine and fertility .Myomectomy can be accomplished by laparotomy, laparoscopy, or hysteroscopy (transvaginal) approaches.

Uterine fibroids have a rich blood supply which may result in intensive bleeding during the myomectomy procedure.This surgical procedure may be associated with substantial morbidity, in particular major blood loss especially in abdominal myomectomy. Fletcher reported that 23% patients undergoing open myomectomy lost over 1000ml of blood. Other studies reported the operative blood loss range between 100 ml and 3000 mls. Blood transfusion can be required in up to 20% of the women during abdominal myomectomy and may require hysterectomy in up to 2% of patient undergoing abdominal myomectomy.

A number of interventions have been introduced to reduce bleeding rate during myomectomy:

1. interventions on uterine arteries as peri cervical mechanical tourniquet, preoperative clamping or embolization of bilateral uterine and/or ovarian arteries (UAE)
2. uterotonics as ergometrine, oxytocin, misoprostol, peri-operative injection of ascorbic acid, or intraoperative vasopressin or terlipressin injection (hormonal tourniquet) into myometrium , or intra-myometrial infiltration of bupivacaine plus epinephrine,
3. myoma dissection techniques as use of laser, electrosurgery and chemical dissectors such as mesna.
4. GnRH analogues reduce haemorrhage during surgery if used for 2-4 months preoperatively. GnRH analogues are expensive and may make removing fibroids difficult because of reduced distinction between capsule and myometrium.

However, these strategies may be associated with some complications, and some of these are ineffective or expensive or require extra steps before the actual procedure.

The Foley catheter, often used as a tourniquet in low resource countries, is cheap and readily available;however, they require intermittent release intraoperatively to prevent the build-up of toxins and tissue ischemia, and may be impracticable to apply sometimes. Once the tourniquet is removed, there is bleeding from the raw myometrium and cavities with the possibility of increased blood loss and blood transfusion. Tourniquet occlusion of uterine and ovarian vessels prior to myomectomy was reported by Kongenyuy et al to have higher efficacy in reducing intraoperative blood loss when compared to other interventions. Mechanical vascular occlusion techniques such as tourniquet or uterine artery embolization, though popular in recent years have significant disadvantages as (i) require additional interventions or a separate procedure during the operation (ii) difficulty of access to the uterine artery with large and laterally placed myomas and (iii) difficulty of placing the tourniquet. In practice,there are instances when application of the tourniquet is impracticable and another method is indicated as in case of significant pelvic adhesions and leiomyoma in the broad ligament, uterine isthmus or cervix.

Medical agents are always an attractive option to arrest haemorrhage. Preoperative Misoprostol, a prostaglandin E1 analogue, was registered in many countries for use in gynaecology and obstetrics. Its popularity in developing countries is accounted by its advantages over other interventions as being inexpensive choice with thermal and light stability and shelf life of several years in tropical conditions. It acts by promoting myometrial contractions and reducing uterine artery blood flow significantly and thus reducing bleeding during myomectomy . Reports on misoprostol use to control blood loss in abdominal myomectomy showed a reduction in intra and post-operative blood loss, surgical time, and post-operative blood transfusion . Misoprostol has advantage of multiple routes of administration as sublingual, oral, rectal or vaginal. The bioavailability curve of rectal and vaginal misoprostol is qualitatively similar although rectal route has longer half-life with lesser side effects than oral route. The peak plasma level of 400 μg of vaginal misoprostol is reached one to two hours after administration and is sustained for four hours, and the side effects are self-limiting . Another advantage of Misoprostol is that it is much cheaper than GnRH analogues; the most popular method for reducing bleeding in myomectomy operation. Another advantage over GnRH analogues is that the effect of GnRH analogues achieved only after an average time of 3 months while misoprostol can be administered an hour before the operation and significantly reduces intra-operative blood loss. Side effects of misoprostol appear within 90 minutes of administration, i.e., while patient is under anaesthesia and are less disturbing in nature such as nausea, vomiting, diarrhea, abdominal pain, fever and chills. Single dose of misoprostol is associated with lower incidence of shivering and hyperpyrexia and with no serious systemic side effects.

Oxytocin is a hormone secreted mainly from the pituitary gland. Its main function is uterine contraction during labour and delivery. Oxytocin is the agent of choice in the prevention of postpartum uterine atony and bleeding. Oxytocin acts directly on the myometrium through the oxytocin receptor(OXTR) and stimulates contractions. Oxytocin affects oxytocin receptors in the myometrium and fibroid tissue, which stimulates synthesis and release of contractile prostaglandins. Increased uterine contractility directly affects uterine vascular structures, decreasing blood supply to the arteries and fibroids. Decreased blood volume in the uterus and constricted uterine vasculature due to uterine contraction and vaso-constrictive effect of oxytocin results in reducing intraoperative blood loss. Oxytocin receptors also exist in the nonpregnant uterus with a 50-100 times lower concentration than in pregnant uterus.The expression of oxytocin receptors have been identified in the endometrium as well as in the microvascular endothelial cells of the myometrium. Further, oxytocin receptors were found to be higher in fibroids than in normal myometrium. Main side effects caused by oxytocin are tachycardia, hyponatremia and hypotension but usually these side effects don't occur with low doses but it should be used cautiously because an intravenous bolus of 10 IU oxytocin could be detrimental to women with heart disease or to women who are hypovolemic.

Nevertheless, oxytocin has a short half-life (4-10 minutes), necessitating continuous intravenous infusion. Moreover, saturation of myometrial oxytocin receptors could reduce its effectiveness, and excessive dosing can lead to coronary-artery contraction and hypotension; additionally, water intoxication can occur owing to its anti-diuretic effects.

Carbetocin is a long-acting synthetic octapeptide analogue of oxytocin(which is a nonapeptide) with agonist properties at the oxytocin receptor. The molecular changes give Carbetocin more stability and avoid early decomposition .Originally, it is an obstetric drug used to control postpartum hemorrhage . In recent times, it has been studied in the reduction of bleeding during myomectomy, but the available data are limited. The pharmacodynamic properties of Carbetocin are comparable to those of endogenous oxytocin.

Carbetocin selectively binds to oxytocin receptors in the smooth muscle of the uterus resulting in rhythmic uterine contractions, increased frequency of existing contractions, and increased uterine tone. During surgery, addition of carbetocin will lead to strong muscle contractions that makes myometrium pale with less bleeding and myoma will become more protruding.

It can be administered as a single-dose injection, either intravenously or intramuscularly or can be given intramyometrial. Intravenously administered Carbetocin has a half-life of approximately 40 minutes, around 4-10 times longer than that reported for oxytocin. Following intramuscular injection, Carbetocin reaches peak plasma concentrations in less than 30 minutes and has 80% bioavailability. Carbetocin onset of action is rapid irrespective of administration route, but duration of action is longer following intramuscular injection as contractions continue for 60 minutes after the intravenous injection and for 120 minutes after the intramuscular administration. The optimal Carbetocin dose (intravenous or intramuscular) is100 μg.

Other methods:

Preoperative uterine embolization decreases blood loss during a myomectomy, however, this option is limited by the accessibility of equipment and by having trained physicians to complete the procedure .

Vasopressin is not a cost-effective choice and there can be associated pulmonary oedema, temporary increase in blood pressure and myocardial infarction with it.

In this study, we will compare the effectiveness of a single preoperative dose of vaginal misoprostol ,intraoperative oxy¬tocin infusion, IV carbetocin and pericervical tourniquet for the reduction of blood loss at the time of abdominal myomectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-40 years.
2. 1-5 symptomatic intramural, submucous or subserous myomas by ultrasound
3. Mean uterine fibroid size of 5-10 cm
4. Presented with abnormal uterine bleeding, dull lower abdominal pain, infertility or recurrent miscarriage and are candidates for abdominal myomectomy.

Exclusion Criteria:

1. History of previous abdominal or pelvic surgery (laparotomy) except Cesarian section.
2. History of pelvic or ovarian endometriosis.
3. History of PID.
4. Patient with pedunculated subserous fibroid.
5. Patients who are candidate for laparoscopic or hysteroscopic myomectomy.
6. Allergy to misoprostol.
7. Hypertension, Diabetes Mellitus, Cardiac and pulmonary diseases.
8. Obesity BMI > 30 kg/m².
9. Anemia Hb < 10 g/dL.
10. Bleeding disorder or use of anticoagulation.
11. Preoperative use of hormonal therapy as GnRH analogues or oral contraceptive pills.
12. Pregnancy.
13. Postmenopausal.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | baseline
  estimated by calculating the sum of canisters containing irrigation fluids and suctioned (ml)blood minus used irrigation solution plus the amount of absorbed blood in used sponges then converting weight with volume of blood loss as [post-operative wet sponge weight in (grams) minus preoperative dry sponge weight (grams) which means 1 ml of blood weighs 1gm].

SECONDARY OUTCOMES:
The need for blood transfusion | baseline
  Number of patients in each group who require transfusion.
Preoperative and postoperative haemoglobin and haematocrit values | 24 hours before and 24 hours after
  (gm/dl) will be measured on 24 hours before and 24 hours after surgery
Perioperative blood pressure and HR | Up to 4 hours postoperative
  Measure blood presure and pulse at start and end of operation and then every hour interval up to first four hours postoperative.
Time of ambulation | within 12 hours postoperative
  interval the operation ended up patient's walking with assistance in hours
Post-operative hospital stay | within 3 days postoperative
  days
Operation time | within 120 minutes
  measured from incision of first myoma to serosal closure of last myoma wound in minutes
Anaesthesia time | with in 120 minutes
  Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ibrahim Aref, professor, Study Chair — Kasr Alainy Cairo University; Soumaya Mohamed AbouElew, professor, Study Chair — Kasr Alainy Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdel-Hafeez M, Elnaggar A, Ali M, Ismail AM, Yacoub M. Rectal misoprostol for myomectomy: A randomised placebo-controlled study. Aust N Z J Obstet Gynaecol. 2015 Aug;55(4):363-8. doi: 10.1111/ajo.12359. Epub 2015 Jul 14. PMID 26174128
- [Background] Atashkhoei S, Fakhari S, Pourfathi H, Bilehjani E, Garabaghi PM, Asiaei A. Effect of oxytocin infusion on reducing the blood loss during abdominal myomectomy: a double-blind randomised controlled trial. BJOG. 2017 Jan;124(2):292-298. doi: 10.1111/1471-0528.14416. Epub 2016 Nov 15. PMID 27862855
- [Background] Farouk H, Shady N (2017) Intravenous Carbetocin to decrease blood loss during open myomectomy: a randomized placebo-controlled study. IJRCOG 7:
- [Background] Gad Allah, S. H., A Wali, A., & Mostafa, S. (2015). Hemostatic effect and postoperative benefits of intramyometrial carbetocin injection during myomectomy: a randomized controlled trial. Evidence Based Women's Health Journal, 5(4), 185-189.
- [Background] Gharabaghi PM, Alizadeh S, Atashkhoye S, Sayyah-Melli M, Jafari- Shobeiri M, Ouladsahebmadarek E, et al. Comparing the Outcomes and Side Effects of Administration of a Single Preoperative Dose of Vaginal Misoprostol With Intraoperative Oxytocin Infusion in Blood Loss During Abdominal Myomectomy. Int J Women's Health Reprod Sci 2017;
- [Background] Kongnyuy EJ, Wiysonge CS. Interventions to reduce haemorrhage during myomectomy for fibroids. Cochrane Database Syst Rev. 2014 Aug 15;2014(8):CD005355. doi: 10.1002/14651858.CD005355.pub5. PMID 25125317
- [Background] Ragab A, Khaiary M, Badawy A. The Use of Single Versus Double Dose of Intra-vaginal Prostaglandin E2 "Misoprostol" prior to Abdominal Myomectomy: A Randomized Controlled Clinical Trial. J Reprod Infertil. 2014 Jul;15(3):152-6. PMID 25202673